CLINICAL TRIAL: NCT06674525
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of SSGJ-626 in Healthy Adult Subjects
Brief Title: Evaluation of 626 in Healthy Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSGJ-626-HV-I-01
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Healthy Subjects (HS)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- 626 Group S1 for subcutaneous injection (Experimental): dose level 1 of 626
  Interventions: Drug: 626; Drug: Placebo
- 626 Group S2 for subcutaneous injection (Experimental): dose level 2 of 626
  Interventions: Drug: 626; Drug: Placebo
- 626 Group S3 for subcutaneous injection (Experimental): dose level 3 of 626
  Interventions: Drug: 626; Drug: Placebo
- 626 Group S4 for subcutaneous injection (Experimental): dose level 4 of 626
  Interventions: Drug: 626; Drug: Placebo
- 626 Group S5 for subcutaneous injection (Experimental): dose level 5 of 626
  Interventions: Drug: 626; Drug: Placebo
- 626 Group S6 for subcutaneous injection (Experimental): dose level 6 of 626
  Interventions: Drug: 626; Drug: Placebo

INTERVENTIONS:
Drug: 626 — Single subcutaneous injection
  Other Names: SSGJ-626
Drug: Placebo — Single subcutaneous injection

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose phase I clinical study to evaluate the safety, tolerability, PK and immunogenicity of SSGJ-626 in healthy adult subjects after single subcutaneous injection.

DETAILED DESCRIPTION:
Six dose groups are planned for dose escalation in this study. Subjects in all dose groups will receive a single subcutaneous injection. Group S1 follows open-labeled, single-arm design, Groups S2 to S6 follow randomized, double-blinded, placebo-control design. Blood samples will be collected for PK, immunogenicity, biomarkers, laboratory tests, etc. according to the study schedule throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand protocol requirements and sign a written ICF.
* Male or female subjects aged 18-45 years when signing the ICF.
* Male subjects with body weight ≥ 50 kg, and female subjects with body weight ≥ 45 kg. Subjects with BMI between 18 and 28 kg/m2.
* Subjects whose test results are normal, or abnormal without clinical significance as determined by the investigator.
* Female subjects with childbearing potential and male subjects (and their female partners) must agree to take highly effective contraceptive measures.

Exclusion Criteria:

* History of severe allergy, or with a history of allergy to the study treatment or related excipients.
* With any clinically significant diseases prior to the screening visit.
* Subjects with positive test results for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibody, anti-human immunodeficiency virus (HIV) antibody.
* History of of significant alcohol abuse.
* History of significant drug abuse.
* Subjects who have positive result for urine nicotine test at screening.
* Pregnant, or nursing females.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 90 days
  Incidence of adverse events will be summarized by SOC and PT for each treatment group, and also be summarized by severity and association with the study treatments.

SECONDARY OUTCOMES:
Cmax | 90 days
  Peak concentration (Cmax) will be calculated.
Tmax | 90 days
  Time to peak concentration (Tmax) will be calculated.
AUC0-last | 90 days
  Area under the concentration-time curve from time 0 to the time point of last measurable concentration post-dose (AUC0-last) will be calculated.
Incidence of Anti-Drug Antibody | 90 days
  Anti-drug antibody (ADA) positive rate and titer will be calculated. Incidence of neutralizing antibody (Nab) if ADA is positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China